CLINICAL TRIAL: NCT02735564
Title: Change in Reward System Activation and Gut Microbiota Following Roux-en-y and Sleeve Gastrectomy for Weight Loss as Compared to a Control- Heads Up Ancillary
Brief Title: Change in Reward System Activation and Gut Microbiota Following RYGB and Sleeve Gastrectomy for Weight Loss vs. Control-Heads Up Ancillary
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Corby K. Martin, Associate Professor, Pennington Biomedical Research Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PBRC 2015-064
Record Dates: First submitted 2016-04-06; First posted 2016-04-12 (Estimated); Last update posted 2020-01-06 (Actual); Status verified 2020-01

CONDITIONS: Bariatric Surgery Candidate
Keywords: Weight Loss; Magnetic Resonance Imaging; gut microbiota
MeSH Terms: conditions — Weight Loss | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- RYGB (Experimental): Bariatric Surgery:Roux-en-y
  Interventions: Procedure: Bariatric Surgery
- SG (Experimental): Bariatric Surgery: Sleeve Gastrectomy
  Interventions: Procedure: Bariatric Surgery
- Control (Placebo Comparator): BMI matched control
  Interventions: Procedure: Bariatric Surgery

INTERVENTIONS:
Procedure: Bariatric Surgery

SUMMARY:
Bariatric surgery is considered an effective long-term intervention for the treatment of obesity and associated complications. While bariatric surgery has been shown to result in a large sustained weight loss, the degree of weight loss and maintenance thereafter varies greatly. The Heads Up Surgical Demonstration Project (Heads Up) is a 5 year project examining weight loss after an intensive medical intervention (IMI) and the 2 most widely used bariatric surgeries (roux-en-y gastric bypass or RYGB and sleeve gastrectomy or SG). Baseline data are collected prior to surgery and follow-up data are collected at 6 months and annually thereafter. A recent meta-analysis revealed that RYGB resulted in greater weight loss and is more effective in resolving obesity related comorbidities than SG, although SG has been shown to result in a reduction of perioperative complications and reoperations1. Full elucidation of the mechanisms leading to variation in success for weight loss interventions is crucial to understanding the most effective and reliable treatments for obesity and associated comorbidities.

ELIGIBILITY:
Inclusion Criteria:

Surgical Groups (RYGB and SG) Inclusion criteria for the two surgery groups (n=16)

* Individuals who qualify for Heads Up and would like to participate in this ancillary study
* Be willing to participate in additional procedures including: 4 brains scans (2 before surgery and 2 after surgery), 2 meal challenges (1 before surgery and 1 after surgery), and 2 microbiota collections (1 before surgery and 1 after surgery).
* Be willing to archive microbiota samples

Control Group:

Inclusion Criteria for the BMI matched control group (n=9):

* Males and females age 21-70 years
* Body Mass Index ≥40 kg/m2 without type 2 diabetes or ≥35 kg/m2 and ≤ 60kg/m² with type 2 diabetes
* Agree to receive frequent contacts from investigators and communicate with program staff for up to 6 months
* Able to give written informed consent
* Able to comply with study procedures

Exclusion Criteria:

* Exclusion Criteria for the two surgery groups (n=16):

  * Unable or unwilling to give informed consent
  * Pregnant or planning on becoming pregnant during the 6 months you participate in the study
  * History or presence of unremoveable metal objects (medical or dental) or electronic devices or other contraindication to MRI scanning.
  * Unwillingness to complete an MRI due to confined space or other related phobias

Exclusion Criteria for the BMI matched control group (n=9):

* Unable or unwilling to give informed consent
* Hospitalization for psychiatric illness or substance use/abuse within the past year
* Diagnosis of schizophrenia, other psychotic disorders, bipolar disorder, or personality disorder as determined by the medical staff
* Travel plans that do not permit participation
* Pregnant or planning on becoming pregnant during the 6 months you participate in the study
* History of prior bariatric surgery, extensive bowel resection, or hiatal hernia repair (unless approved by the medical staff)
* History of eating disorder such as anorexia nervosa, bulimia, or binge eating (unless approved by program staff)
* Current major depressive episode or history of suicidal behaviors
* Severe congestive heart failure (NYHA class III, IV)
* Second degree or greater heart block
* Other medical, psychiatric, or behavioral limitations that in the judgement of the investigator may interfere with program participation or the ability to follow the intervention protocol
* History or presence of unremoveable metal objects (medical or dental) or electronic devices or other contraindication to MRI scanning.
* Unwillingness to complete an MRI due to confined space or other related phobias

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Neural reward sensitivity | baseline, 6 months
  Investigate change in reward activation patterns in the brain in response to food cues using fMRI.
gut microbiota | baseline, 6 months
  Determine if gut microbiota, as analyzed via stool sample collection, changes from baseline (prior to surgery) to 6 months follow-up (post-surgery) among the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Keely Hawkins, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No